



## Identify the prosthesis users' necessities concerning their devices.

VITÓRIA, BRASIL 6 DE NOVEMBRO 2023





| Priginal | |
|---|---|
| Original Primary Outcome<br>Measures ICMJE | Number of patients that have an unconformity with the weight of the device and which functional characteristics they would improve their devices s concerning their devices. |
| Current Secondary Outcome<br>Measures ICMJE | - |
| Brief Summary (5000 Ch) | Despite many advances in prosthesis development, there are still some areas that need to be improved. One of them is the weight of the devices which could cause muscular fatigue in long-term use of the prosthesis and even abandonment. This study aims to identify the desired improvements in prosthetic devices from the perspective of the users, therapists, and relatives. That would be done through two kinds of questionnaires about technology acceptance. |
| Detailed Description (32000<br>Ch) | The World Health Organization (WHO) estimates that around 1.3 billion people experience significant disability. One of the actual challenges is facilitating and breaking the barriers of persons with disabilities. Assistance technology supports inclusion and participation, principally for people with disabilities. |
| | In Brazil, the DATASUS estimated that around 57802 amputations (one kind of disability) were performed in 2022. Prostheses are assistive devices that aim to mitigate the psychological impact of missing a member and help in activities of daily life (ADL). One kind of prosthesis is electrically powered, which uses electrical components to actuate the device and is commonly controlled by body signals such as surface electromyography (sEMG). Despite many advances in prosthesis development, some areas need to be improved such as weight, size, ergonomic design, etc. of the devices which could cause muscular fatigue in long-term use of the prosthesis and even abandonment. |
| | This study aims to identify the aspects that cause major discomfort in upper limb prosthesis users. Also, recognize in which activities of daily life, the prosthesis is involved. That information will be used to improve the design of an upper limb prosthesis. |
| Study Type ICMJE | Observational, qualitative-quantitative study |
| Study Phase ICMJE | Waiting for the approval to contact the prosthesis users |
| Study Design ICMJE | The study is grounded on a non-invasive protocol, which investigates the necessities in the design of the upper limb prosthesis from the users', relatives', and therapist's perspectives. |
| Condition ICMJE | Upper limb amputees |
| Intervention ICMJE | For the execution, three kinds of questionnaires about technology acceptance will be used. In the first questionnaire, which is for prosthesis users, there will be 15 questions to identify what kind of activities the person uses the prosthesis, how much is the use time and what is the main problem with the device. In the second and third questionnaires, |





| | between 8 and | the therapist and relatives respectively, there will be 9 questions to analyze which device characteristics, they e major discomfort during the use and could be improved. |
|---|---|---|
| Study Arms ICMJE | Arm Prosthesis Users Therapists Relatives | Description 30 participants, aged between 18 and 60, will be part of the study. It is necessary that the users have at least 6 months of experience using upper limb prostheses. 10 therapists that have experience working with prostheses. 30 of the prosthesis users' relatives who live with the person and see the daily difficulties of using |
| | | the device, |





| Publications * |
|----------------|





| Recruitment Information | |
|---|---|
| Recruitment Status ICMJE | Enrolling by invitation |
| Actual Enrollment ICMJE | Participants will be selected from a predetermined population |
| Original Actual<br>Enrollment ICMJE | |
| Actual Study Completion Date ICMJE | September 2024 |
| Actual Primary Completion<br>Date | September 2024 |
| Eligibility Criteria ICMJE | Prosthesis users with at least 6 months of device use. A therapist with experience in working with amputees. Relatives of the prosthesis users. |
| Sex/Gender ICMJE | Mixed |
| Ages ICMJE | 18 to 60 years |
| Accepts Healthy<br>Volunteers ICMJE | - |
| Contacts ICMJE | Laura Vanesa De Arco Barraza |